CLINICAL TRIAL: NCT06197191
Title: Holter and ECG Changes After Trancatheter Closure Of ASD In Children
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abdelgalil, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-04-12
Record Dates: First submitted 2022-04-17; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: ASD II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fukuda Denshi Cardimax ECG device model FCP-7101 — ecg and holter will be done one day before and one day after then after 1,6,12 month after transcatheter closure of ASD
  Other Names: Holter ECG mortara H3+

SUMMARY:
Atrial septal defects (ASD) account for 10% of all congenital heart defects . Hemodynamic consequences of an ASD are dilatation of the right atrium and right ventricle (RV) because of the volume overload due to the left-to-right shunt through the ASD.For several decades, surgical closure has been considered the standard method of repairing a secundum ASD . Surgical repair, albeit enjoying a high success rate, negligible mortality, and good long-term outcome, is associated with morbidity, discomfort, and thoracotomy scars. That is why the transcatheter closure of the ASD has more recently become an alternative to the surgical procedure . During the last decade , ASD device closure , has finally replaced surgical ASD repair in most patients as the standard method of repair for the secundum ASD Cardiac arrhythmias and right chamber enlargement are well known long-term sequelae of atrial septal defect (ASD) . Therefore, many authors suggest ASD closure before adulthood . Classical ECG findings for a significant ASD are prolongation of the PR interval, prolongation of the QRS duration and right axis deviation of the QRS .

Percutaneous ASD closure is an ideal situation to study changes of RV dimensions and their impact on ECG as interferences from cardiopulmonary bypass, cardiac incisions and sutures on the right atrium and on the interatrial septum are excluded

ELIGIBILITY:
Inclusion Criteria:

* All children under the age of 18 years diagnosed with ASD , that will undergo transcatheter secundum ASD device closure during the period of the study .

Exclusion Criteria:

* Failure to obtain informed consent .

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: - All children under the age of 18 years diagnosed with ASD , that will undergo transcatheter secundum ASD device closure during the period of the study .
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
ECG Changes after transcatheter closure of ASD | one year
  ECG will be done one day before and one day after then after 1,6,12 month of ASD closure , determination of the following variables ; heart rate, QRS axis, PR interval , QRS duration and the QT interval . Interpretation of every ECG paper was done using specific centile tables for normal values of ECG waves and intervals according to age . ECG will be examined for any abnormal rhythm (heart block, ectopics ,supraventricular or ventricular tachycardia) .
HOLTER ECG Changes after transcatheter closure of ASD | one year
  Six channel Holter ECG will be used for recording the day before , the day after the procedure then repeated at 1m,6m and 12m . the recordings will be used for evaluation of mean HR, Mean QTC interval duration .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Celiker A, Ozkutlu S, Karagoz T, Ayabakan C, Bilgic A. Transcatheter closure of interatrial communications with Amplatzer device: results, unfulfilled attempts and special considerations in children and adolescents. Anadolu Kardiyol Derg. 2005 Sep;5(3):159-64. PMID 16140642
- [Background] Masura J, Gavora P, Podnar T. Long-term outcome of transcatheter secundum-type atrial septal defect closure using Amplatzer septal occluders. J Am Coll Cardiol. 2005 Feb 15;45(4):505-7. doi: 10.1016/j.jacc.2004.10.066. PMID 15708695
- [Background] Peters B, Ewert P, Schubert S, Abdul-Khaliq H, Schmitt B, Nagdyman N, Berger F. Self-fabricated fenestrated Amplatzer occluders for transcatheter closure of atrial septal defect in patients with left ventricular restriction: midterm results. Clin Res Cardiol. 2006 Feb;95(2):88-92. doi: 10.1007/s00392-006-0329-3. Epub 2006 Jan 16. PMID 16598516